CLINICAL TRIAL: NCT03615248
Title: Effectiveness of a Mobile Health Intervention in Improving the Technique of Inhaled Medications Among Children With Asthma: A Pilot Study
Brief Title: Effectiveness of a Mobile Health Intervention in Improving the Technique of Inhaled Medications Among Children With Asthma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Mary Jane Smith, Assistant Professor of Pediatrics, Memorial University of Newfoundland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MemorialUN001
Record Dates: First submitted 2018-07-18; First posted 2018-08-03 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Asthma; Asthma in Children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Arm - (Experimental): 30 Subjects will be approached in Asthma Clinics at the Janeway Children's Health and Rehabilitation Centre by the research nurse, and if selected to the study, will use the BreatheSuite device for 3-6 months.
  Inclusion criteria: Age 10-18, diagnosis of asthma by the pediatrician, regular access to a smartphone, parental consent, ongoing need for regular use of a medication delivered by metered dose inhaler as deemed by the pediatrician, ability to demonstrate proper technique of metered dose inhaler use in the clinic while supervised by research nurse or pediatrician without parent or caregiver intervention;
  Interventions: Device: BreatheSuite

INTERVENTIONS:
Device: BreatheSuite — BreatheSuite (patent pending) is a device and mobile application developed by Mr. Brett Vokey, an engineering student at Memorial University of Newfoundland. BreatheSuite has been recognized by numerous provincial competitions, featured at the Eastern Health Innovation Showcase, and was recently selected as a finalist for the New York Health Innovation Challenge.
  This device attaches to metered dose inhalers and it can determine if:
  1. the dose was given,
  2. the metered dose inhaler was properly shaken,
  3. the metered dose inhaler is properly aligned,
  4. the flow of medication is appropriate and
  5. there is no accidental exhalation into the inhaler.

SUMMARY:
In this trial, the investigators aim to determine if a new mobile health intervention (BreatheSuite) can increase inhaler technique and adherence amongst participants aged 10-18. See the below detailed description for more information.

DETAILED DESCRIPTION:
Improper inhaler technique can significantly affect the amount of medication reaching the lungs and patients with the incorrect technique are likely to have poorly controlled asthma and more emergency department visits. Studies have shown that up to 92% of children demonstrate poor inhaler technique. A systematic review of errors in inhaler technique showed that most errors were in coordination, speed or depth of inspiration, and no post inhalation breath-hold.

BreatheSuite (patent pending) is a device and mobile application developed by Mr. Brett Vokey, an engineering student at Memorial University of Newfoundland. BreatheSuite has been recognized by numerous provincial competitions, featured at the Eastern Health Innovation Showcase, and was recently selected as a finalist for the New York Health Innovation Challenge.

This device attaches to metered dose inhalers and it can determine if:

1. the dose was given,
2. the metered dose inhaler was properly shaken,
3. the metered dose inhaler is properly aligned,
4. the flow of medication is appropriate, and
5. there is no accidental exhalation into the inhaler.

All of this information is transmitted to the BreatheSuite mobile application, which is then available to the user. The user will get technique correcting advice via push notifications as well as by accessing the mobile application directly. The healthcare professional can look at the data to determine where more education can be given and tailor treatment to the individual.

Similar to that done of a study by Ronmark et al, inhaler technique scores are computed from 0-100%, with each of the five technique steps mentioned above are given one of three values: 20 (Perfect Score for Technique Step), 10 (partially correct step) or 0 (not correct at all). Thus, the technique scores are varied from 0-100 in increments of 10.

One downfall of many metered dose inhalers is that they do not include a dose indicator. The patient can not know how many doses are remaining. The number of doses in each metered dose inhaler is clearly labelled on the canister. However, if patients are not keeping track in their asthma logbook, or elsewhere, they may not know when their device is empty. This downfall can lead to omitted doses and poor control. BreatheSuite's ability in monitoring doses has the potential to enhance medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-18,
* diagnosis of asthma by the pediatrician,
* regular access to a smartphone,
* parental consent,
* ongoing need for regular use of a medication delivered by metered dose inhaler as deemed by the pediatrician,
* ability to demonstrate proper technique of metered dose inhaler use in the clinic while supervised by Asthma Nurse or pediatrician without parent or caregiver intervention

Exclusion Criteria:

* Children 9 or under.
* Individuals not using a metered dose inhaler.
* Individuals without a smartphone.
* Individuals taking part in another drug/device study at this time
* Individuals who have finished another drug/device study in the last 30 days

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Does the given mobile health intervention improve inhaler technique in children aged 10-18? | 3-6 Months
  Detailed outcome measures include:
  To compare the metered dose inhaler technique before and after use of BreatheSuite.This device attaches to metered dose inhalers and it can determine if:
  1. the dose was given,
  2. the metered dose inhaler was properly shaken,
  3. the metered dose inhaler is properly aligned, and
  4. the flow of medication is appropriate.
  5. there is no accidental exhalation into the inhaler.
  Similar to that done of a study by Ronmark et al, inhaler technique scores are computed from 0-100%, with each of the five technique steps mentioned above are given one of three values: 20 (Perfect Score for Technique Step), 10 (partially correct step) or 0 (not correct at all). Thus, the technique scores are varied from 0-100 in increments of 10.

SECONDARY OUTCOMES:
To compare the Asthma Control Questionnaire scores before and after use of BreathSuite | 3-6 months
  Asthma Control Questionnaire is a validated questionnaire which assesses asthma control over the previous week. It will be administered at the beginning of the study and upon study completion 3-6 months later

OTHER OUTCOMES:
To compare patient satisfaction between BreatheSuite and the logbook | 3-6 months
  At the end of the study a short Exit Survey has will be administered which asks subjects about their experience including whether they prefer using Breathesuite to track their inhaler use or an asthma logbook.
To assess patient satisfaction with BreatheSuite | 3-6 months
  A the end of the study a short Exit Survey will be administered which asks subjects their level of satisfaction with Breathesuite.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jane Smith, MD, Principal Investigator — Memorial University of Newfoundland
Locations (1):
- Memorial University of Newfoundland, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Sickle D, Magzamen S, Truelove S, Morrison T. Remote monitoring of inhaled bronchodilator use and weekly feedback about asthma management: an open-group, short-term pilot study of the impact on asthma control. PLoS One. 2013;8(2):e55335. doi: 10.1371/journal.pone.0055335. Epub 2013 Feb 27. PMID 23460785
- [Background] Al-Jahdali H, Ahmed A, Al-Harbi A, Khan M, Baharoon S, Bin Salih S, Halwani R, Al-Muhsen S. Improper inhaler technique is associated with poor asthma control and frequent emergency department visits. Allergy Asthma Clin Immunol. 2013 Mar 6;9(1):8. doi: 10.1186/1710-1492-9-8. PMID 23510684
- [Background] Burkhart PV, Rayens MK, Bowman RK. An evaluation of children's metered-dose inhaler technique for asthma medications. Nurs Clin North Am. 2005 Mar;40(1):167-82. doi: 10.1016/j.cnur.2004.08.010. PMID 15733954
- [Background] Sleath B, Ayala GX, Gillette C, Williams D, Davis S, Tudor G, Yeatts K, Washington D. Provider demonstration and assessment of child device technique during pediatric asthma visits. Pediatrics. 2011 Apr;127(4):642-8. doi: 10.1542/peds.2010-1206. Epub 2011 Mar 28. PMID 21444594
- [Background] Ronmark E, Jogi R, Lindqvist A, Haugen T, Meren M, Loit HM, Sairanen U, Sandahl A, Lundback B. Correct use of three powder inhalers: comparison between Diskus, Turbuhaler, and Easyhaler. J Asthma. 2005 Apr;42(3):173-8. PMID 15962873